CLINICAL TRIAL: NCT01912534
Title: Valsartan for Attenuating Disease Evolution In Early Sarcomeric HCM
Acronym: VANISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VANISH; 5P50HL112349 (NIH)
Record Dates: First submitted 2013-06-05; First posted 2013-07-31 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2020-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Sarcomere Mutations
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): Subjects who tolerate active run-in and titration to target dose of valsartan will then undergo stratified randomization and begin blinded treatment with valsartan or matched placebo on maximal tolerated dose, according to their assigned treatment group. Treatment will continue for 2 years.
  Interventions: Drug: Valsartan; Drug: Placebo
- Placebo (Placebo Comparator): Subjects who tolerate active run-in and titration to target dose of valsartan will then undergo stratified randomization and begin blinded treatment with valsartan or matched placebo on maximal tolerated dose, according to their assigned treatment group. Treatment will continue for 2 years.
  Interventions: Drug: Valsartan; Drug: Placebo

INTERVENTIONS:
Drug: Valsartan — 40, 80 and 160 mg tablets of Valsartan
  Other Names: Diovan
Drug: Placebo — During Active Run-In, all patients take Valsartan. During maintenance, all patients are randomized to valsartan or placebo
  Other Names: Matching Placebo pills

SUMMARY:
The purpose of this trial is to determine whether treatment with valsartan will have beneficial effect in early hypertrophic cardiomyopathy (HCM) by assessing many domains that reflect myocardial structure, function and biochemistry.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled Phase II, randomized clinical trial to assess the safety and efficacy of valsartan in attenuating disease evolution in early HCM. Sarcomere mutation carriers with asymptomatic or mildly symptomatic overt disease (NYHA class I-II), and mutation carriers without left ventricular hypertrophy (LVH) will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have a Pathogenic or Likely Pathogenic HCM Sarcomere Mutation

a. The following categories of mutations are considered acceptable for subjects who have previously undergone clinical genetic testing. If results are ambiguous, they will be reviewed by the Clinical Coordinating Center to determine eligibility.

* Laboratory for Molecular Medicine (Pathogenic, Likely Pathogenic)
* Transgenomics/ PGXHealth (Class I)
* GeneDx (Disease causing; Variant; likely disease-causing; Published, disease-causing mutation; Novel, likely disease-causing, mutation)
* Correlagen (Associated; Probably Associated)

Group 1 (Overt HCM Cohort)

1. LV wall thickness ≥12 mm and ≤25 mm or z score ≥3 and ≤18 as determined by rapid assessment by the echocardiographic core laboratory
2. NYHA functional class I or II; no perceived or only slight limitations in physical activities
3. No resting or provokable LV obstruction (peak gradient ≤ 30 mmHg) on clinically-obtained Exercise Tolerance Test (ETT)-echo within the past 24 months or transthoracic echo with Valsalva maneuver within the past 12 months
4. Age 8-45 years
5. Able to attend follow-up appointments, complete all study assessments, and provide written informed consent

Group 2 (Preclinical HCM Cohort (G+/LVH-))

1. LV Wall Thickness <12 mm and z score <3 , as determined by rapid assessment by the echocardiographic core laboratory
2. Age 10-25 years
3. E' z score ≤ -1.5 OR ECG abnormalities other than NSSTW changes (Q waves, T wave inversion, repolarization changes) OR LV wall thickness z-score 1.5-2.9 combined with LV thickness to dimension ratio ≥0.19 (as determined by rapid assessment by the echocardiographic core laboratory)
4. Able to attend follow-up appointments, complete all study assessments, and provide written informed consent

Subject Exclusion Criteria

1. Contraindication to angiotensin receptor blocker (ARB) administration, including impaired renal function, hyperkalemia (serum K>5.0 mmol/L), prior history of angioedema
2. Medical conditions associated with increased collagen turnover that may confound interpretation of biomarkers of collagen synthesis (liver, pulmonary or renal fibrosis, inflammatory states, cancer, trauma or surgery within 6 months of enrollment)
3. Concomitant use of Spironolactone, Lithium, or Aliskiren, ARB or ACE-inhibitors. If these drugs are in active use but not necessary for medical care, they may be discontinued and baseline studies can be performed after a 2-week washout period.
4. Pregnant or breastfeeding females - Females of childbearing potential with no effective contraceptive method (including abstinence)
5. Uncontrolled systemic HTN [persistent SBP>160 and/or DBP>90 in adult or equivalent in children (e.g., SBP>99th or DBP>95th percentile for sex, age, and height centile based on the American Academy of Pediatrics normal values)]
6. Obstructive physiology, defined by resting, Valsalva-provoked or exercise-induced gradient >30mmHg within the past 24 months
7. Prior septal myectomy or alcohol septal ablation
8. Known, suspected, or symptomatic coronary artery disease or evidence of prior myocardial infarction based on symptoms or cardiac imaging
9. More than mild valvular heart disease or clinically significant congenital heart disease. Allowable conditions include bicuspid aortic valve without clinically significant stenosis or regurgitation; spontaneously closed ventricular septal defects; patent foramen ovale, small (≤ 2 mm) restrictive ventricular septal defects with normal ventricular size, and other minor defects that are considered allowable after [review and consensus by participating pediatric cardiologists, overall study PI and] adjudication by the echocardiographic core laboratory.
10. Left ventricular ejection fraction (LVEF) <55%
11. Concomitant medical conditions that would preclude performance of or confound interpretation of echocardiography, exercise testing, or CMR (e.g., renal insufficiency, lung disease, orthopedic/rheumatologic conditions, atrial fibrillation)
12. Secondary prevention implantable cardioverter-defibrillator device (ICD; primary prevention ICDs without a history of appropriate therapy, including shock or ATP, are allowable).
13. Prior treatment or hospitalization for symptomatic heart failure
14. Participation in a clinical trial (except observational studies) involving investigational medications within the previous 30 days.

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 211 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Composite z-score | 2 years
  Composite z-score which is the average of 9 change-scores of: serum NTproBNP, serum high-sensitivity cardiac troponin, left ventricular (LV) mass, left atrial (LA) volume, LV end diastolic volume, LV end systolic volume, maximal LV wall thickness, echo E' velocity, echo S' velocity

SECONDARY OUTCOMES:
z-score serum NTproBNP | 2 years
  Z-score for the 2 year change for serum NTproBNP
z-score high sensitivity cardiac troponin | 2 years
  Z-score for the 2 year change for high-sensitivity cardiac troponin
z-score LV mass | 2 years
  Z-score for the 2 year change in LV Mass
z-score LA volume | 2 years
  Z-score for the 2 year change in LA Volume
z-score LV end diastolic volume | 2 years
  Z-score for the 2 year change in LV end diastolic volume
z-score LV end systolic volume | 2 years
  Z-score for the 2 year change in LV end systolic volume
z-score maximal LV wall thickness | 2 years
  Z-score for the 2 year change in Maximal LV wall thickness
z-score echo E' velocity | 2 years
  Z-score for the 2 year change in echo E' velocity
z-score echo S' velocity | 2 years
  Z-score for the 2 year change in echo S' velocity
Binary indicator of success or failure | 2 years
  Success defined as an improvement at 2 years in any of the following: serum NTproBNP, serum high-sensitivity troponin, LV Mass, LA Volume, LV end diastolic volume, LV end systolic volume, Maximal LV wall thickness, echo E' velocity, or echo S' velocity

OTHER OUTCOMES:
Safety of valsartan as assessed by incidence of adverse events | 2 years
  Safety of valsartan as assessed by incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y. Ho, MD, Principal Investigator — Brigham and Women's Hospital
Locations (15):
- United States (13):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School Medicine, St Louis, Missouri
  - Cinncinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Sick Kids, Toronto, Ontario

REFERENCES:
- [Derived] Topriceanu CC, Vissing CR, Axelsson Raja A, Day SM, Russell MW, Zahka K, Pereira AC, Colan SD, Murphy AM, Canter C, Bach RG, Wheeler MT, Rossano JW, Owens AT, Mestroni L, Taylor MRG, Moon JC, Captur G, Patel AR, Wilmot I, Soslow JH, Becker JR, Seidman CE, Lakdawala NK, Bundgaard H, Tahir UA, Ho CY. Proteomic Analysis of Valsartan for Attenuating Disease Evolution in Early Sarcomeric Hypertrophic Cardiomyopathy (VANISH) Clinical Trial. Circ Heart Fail. 2025 Jun;18(6):e012393. doi: 10.1161/CIRCHEARTFAILURE.124.012393. Epub 2025 May 9. PMID 40340372
- [Derived] Ostrominski JW, Claggett BL, Jerosch-Herold M, Raja AA, Day SM, Russell MW, Zahka K, Pereira AC, Colan SD, Murphy AM, Canter C, Bach RG, Wheeler MT, Rossano JW, Owens AT, Mestroni L, Taylor MRG, Patel AR, Wilmot I, Soslow JH, Becker JR, Lakdawala NK, Bundgaard H, Vargas JD, Ho CY; Valsartan for Attenuating Disease Evolution in Early Sarcomeric Hypertrophic Cardiomyopathy (VANISH) Investigators. Valsartan and Cardiac Remodeling in Early-Stage Hypertrophic Cardiomyopathy: The VANISH Randomized Clinical Trial Cardiac Magnetic Resonance Substudy. JAMA Cardiol. 2025 Jun 1;10(6):617-623. doi: 10.1001/jamacardio.2024.5677. PMID 40042824
- [Derived] Ireland CG, Burstein DS, Day SM, Axelsson Raja A, Russell MW, Zahka KG, Pereira A, Canter CE, Bach RG, Wheeler MT, Rossano JW, Owens AT, Bundgaard H, Mestroni L, Taylor MRG, Patel AR, Wilmot I, Soslow JH, Becker JR, Giverts I, Orav EJ, Claggett B, Lin KY, Ho CY. Quality of Life and Exercise Capacity in Early Stage and Subclinical Hypertrophic Cardiomyopathy: A Secondary Analysis of the VANISH Trial. Circ Heart Fail. 2024 Aug;17(8):e011663. doi: 10.1161/CIRCHEARTFAILURE.124.011663. Epub 2024 Aug 1. PMID 39087355
- [Derived] Vissing CR, Axelsson Raja A, Day SM, Russell MW, Zahka K, Lever HM, Pereira AC, Colan SD, Margossian R, Murphy AM, Canter C, Bach RG, Wheeler MT, Rossano JW, Owens AT, Benson L, Mestroni L, Taylor MRG, Patel AR, Wilmot I, Thrush P, Soslow JH, Becker JR, Seidman CE, Lakdawala NK, Cirino AL, McMurray JJV, MacRae CA, Solomon SD, Bundgaard H, Orav EJ, Ho CY; Valsartan for Attenuating Disease Evolution in Early Sarcomeric Hypertrophic Cardiomyopathy (VANISH) Investigators. Cardiac Remodeling in Subclinical Hypertrophic Cardiomyopathy: The VANISH Randomized Clinical Trial. JAMA Cardiol. 2023 Nov 1;8(11):1083-1088. doi: 10.1001/jamacardio.2023.2808. PMID 37672268
- [Derived] Ho CY, Day SM, Axelsson A, Russell MW, Zahka K, Lever HM, Pereira AC, Colan SD, Margossian R, Murphy AM, Canter C, Bach RG, Wheeler MT, Rossano JW, Owens AT, Bundgaard H, Benson L, Mestroni L, Taylor MRG, Patel AR, Wilmot I, Thrush P, Vargas JD, Soslow JH, Becker JR, Seidman CE, Lakdawala NK, Cirino AL; VANISH Investigators; Burns KM, McMurray JJV, MacRae CA, Solomon SD, Orav EJ, Braunwald E. Valsartan in early-stage hypertrophic cardiomyopathy: a randomized phase 2 trial. Nat Med. 2021 Oct;27(10):1818-1824. doi: 10.1038/s41591-021-01505-4. Epub 2021 Sep 23. PMID 34556856
- [Derived] Axelsson Raja A, Shi L, Day SM, Russell M, Zahka K, Lever H, Colan SD, Margossian R, Hall EK, Becker J, Jefferies JL, Patel AR, Choudhury L, Murphy AM, Canter C, Bach R, Taylor M, Mestroni L, Wheeler MT, Benson L, Owens AT, Rossano J, Lin KY, Pahl E, Pereira AC, Bundgaard H, Lewis GD, Vargas JD, Cirino AL, McMurray JJV, MacRae CA, Solomon SD, Orav EJ, Braunwald E, Ho CY. Baseline Characteristics of the VANISH Cohort. Circ Heart Fail. 2019 Dec;12(12):e006231. doi: 10.1161/CIRCHEARTFAILURE.119.006231. Epub 2019 Dec 9. PMID 31813281
- [Derived] Lee TM, Hsu DT, Kantor P, Towbin JA, Ware SM, Colan SD, Chung WK, Jefferies JL, Rossano JW, Castleberry CD, Addonizio LJ, Lal AK, Lamour JM, Miller EM, Thrush PT, Czachor JD, Razoky H, Hill A, Lipshultz SE. Pediatric Cardiomyopathies. Circ Res. 2017 Sep 15;121(7):855-873. doi: 10.1161/CIRCRESAHA.116.309386. PMID 28912187